CLINICAL TRIAL: NCT07351591
Title: Patient-Derived Tumor Organoid Drug Sensitivity Testing to Guide Treatment Selection in Patients With Unresectable Biliary Tract Cancers: A Prospective, Non-randomized, Open-label, Single-Center Phase II Clinical Trial
Brief Title: A Phase II Trial of Organoid Drug Sensitivity Testing to Guide Therapy in Unresectable Biliary Tract Cancers
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, Shen Feng, Professor, Eastern Hepatobiliary Surgery Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EHBHKY2025-H033-P001
Record Dates: First submitted 2026-01-10; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Advanced Biliary Tract Cancer(BTC)
Keywords: organoid; drug-sensitive test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Physician's Choice Group：According to empirical and clinical practice
  Interventions: Drug: Organoid Drug Sensitivity Testing-Guided Therapy

INTERVENTIONS:
Drug: Organoid Drug Sensitivity Testing-Guided Therapy — Fresh tumor tissue from resection is used to establish and culture patient-derived organoids. Successful organoids undergo drug sensitivity testing against a predefined panel of drugs (Gemcitabine + Cisplatin,Gemcitabine + Oxaliplatin,Durvalumab + Gemcitabine + Cisplatin,Pembrolizumab + Gemcitabine + Cisplatin,Toripalimab + Lenvatinib + Gemcitabine + Oxaliplatin). The most effective drug(s), based on IC50 and AUC values, are recommended for treatment

SUMMARY:
This is a prospective, non-randomized, open-label, single-center phase II clinical trial. It aims to evaluate the efficacy and feasibility of using patient-derived tumor organoid drug sensitivity testing (ODST) to guide personalized systemic therapy for patients with unresectable biliary tract cancers (BTC). A total of 88 eligible patients will be enrolled and grouped based on patient preference into either the ODST-guided group or the control group (standard therapy). Tumor tissues obtained via biopsy will be used to establish organoid cultures. Drug sensitivity testing will be performed on a panel of approved regimens (including GC, GEMOX, Durvalumab+GC, Pembrolizumab+GC, and Toripalimab+Lenvatinib+GEMOX) to identify the most effective treatment. Patients for whom organoid testing fails or results are unavailable within one month will receive standard therapy. The primary endpoints are Objective Response Rate (ORR) and Progression-Free Survival (PFS). Secondary endpoints include Overall Survival (OS) and safety profiles. The study seeks to provide a novel, personalized treatment strategy to improve outcomes for patients with advanced BTC.

DETAILED DESCRIPTION:
1. Study Design:

   This is a single-center, prospective, non-randomized, open-label, controlled phase II clinical trial conducted at the Third Affiliated Hospital of Naval Medical University.
2. Study Population:

   The study will enroll 88 adult patients (aged 18-70) with unresectable biliary tract cancers, confirmed per NCCN guidelines. Participants must have an ECOG performance status of 0-1, a life expectancy of >12 weeks, and adequate organ function.
3. Interventions:

   Organoid Drug Sensitivity Testing (ODST) Group: Tumor tissue from biopsies is used to establish patient-derived organoids. Successful organoids undergo drug sensitivity testing against a predefined panel of regimens. The most effective drug(s), based on IC50 and AUC values, are recommended for treatment.

   Control Group (Standard Therapy): Patients receive physician's choice of standard systemic therapy, including GC, GEMOX, or other approved regimens.
4. Study Endpoints:

   Primary Endpoints:

   Objective Response Rate (ORR) as assessed by RECIST 1.1.

   Progression-Free Survival (PFS).

   Secondary Endpoints:

   Overall Survival (OS).

   Safety and tolerability, assessed by the incidence and severity of adverse events (AEs, SAEs) according to NCI CTCAE v5.0.
5. Follow-up:

   Patients will be followed regularly with imaging assessments every 42 days (±3 days) for the first 48 weeks, and every 63 days (±3 days) thereafter. Laboratory tests and clinical evaluations will be conducted to monitor treatment response and adverse events until death, withdrawal of consent, or study termination.
6. Statistical Analysis:

Sample size was calculated based on an assumed improvement in ORR from 26.7% in the control group to 66.7% in the ODST-guided group (α=0.05, power=80%, 1:1 allocation, 10% dropout rate). Statistical analyses will be performed using SAS, with descriptive statistics for safety and efficacy analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged between 18 and 70 years (inclusive).
2. Diagnosis of biliary tract malignancy confirmed according to the NCCN Clinical Practice Guidelines.
3. The subject or their legal guardian understands and voluntarily signs the Informed Consent Form, and is willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures as required by the protocol.
4. The subject is not a candidate for curative resection, transplantation, or local ablation therapy. This includes patients with recurrent disease after prior radical therapy who are not eligible for further curative resection or ablation.
5. Life expectancy of at least 12 weeks.
6. No radiotherapy within 12 weeks prior to the first dose of the study drug.
7. Liver function classified as Child-Pugh Class A or Class B with a score of 7.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
9. Adequate organ and bone marrow function, defined by the following laboratory values within 7 days prior to randomization (without receiving any blood transfusions, hematopoietic growth factors, albumin, or other corrective drugs within 14 days prior to the laboratory tests):

   9.1. Hematological:
   * Absolute Neutrophil Count (ANC) ≥ 1.5 × 10⁹/L
   * Platelet count (PLT) ≥ 75 × 10⁹/L
   * Hemoglobin (HGB) ≥ 9.0 g/dL 9.2. Hepatic:
   * Total Bilirubin (TBIL) ≤ 3 × Upper Limit of Normal (ULN)
   * Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), and Alkaline Phosphatase (ALP) ≤ 5 × ULN
   * Serum Albumin ≥ 28 g/L 9.3. Renal:
   * Serum Creatinine (Cr) ≤ 1.5 × ULN or Creatinine Clearance (CCr) ≥ 50 mL/min (calculated using the Cockcroft-Gault formula)
   * Urinalysis indicates urine protein < 2+; if baseline urinalysis shows urine protein ≥ 2+, a 24-hour urine collection must demonstrate 24-hour urine protein quantification < 1 g.

   9.4. Coagulation:

   * International Normalized Ratio (INR) and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN
10. For women of childbearing potential (WOCBP), a negative urine or serum pregnancy test must be confirmed within 3 days prior to the first dose of study drug (Cycle 1, Day 1). If a urine test is inconclusive, a serum pregnancy test is required. WOCBP and male subjects must agree to use adequate contraception during the observation period and for at least 8 weeks after the last dose of the study drug. A woman is considered not of childbearing potential if she is postmenopausal (≥1 year without menses) or has undergone surgical sterilization (bilateral oophorectomy, hysterectomy, or bilateral tubal ligation). Subjects (both male and female) with risk of pregnancy must use highly effective contraception (with a failure rate of <1% per year) during the entire treatment period and for 120 days after the last dose of the study drug (or 180 days after the last dose of chemotherapy agents).

Exclusion Criteria:

1. Uncorrectable coagulopathy or individuals with a significant bleeding tendency.
2. Evidence of any concurrent malignant disease.
3. Diagnosis of another malignancy within 3 years prior to the first dose, except for radically treated cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, and/or carcinoma in situ that has undergone curative resection.
4. Patients requiring long-term anticoagulant or antiplatelet therapy that cannot be discontinued.
5. Presence of hepatic encephalopathy or refractory pleural effusion/ascites requiring therapeutic intervention.
6. Other anti-tumor or systemic therapies within 2 weeks prior to enrollment:

   * Treatment with Chinese herbal medicine with demonstrated anti-tumor properties.
   * Treatment with Chinese herbal medicine with anti-tumor indications or drugs with immunomodulatory effects (including thymosin, interferon, interleukin), except for localized use to control pleural effusion.
7. History of systemic treatment for active autoimmune disease or ongoing immunosuppressive therapy:

   * Active autoimmune disease requiring systemic treatment (e.g., disease-modifying drugs, corticosteroids, or immunosuppressants) within 2 years prior to the first dose. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement for adrenal or pituitary insufficiency) is not considered systemic treatment.
   * Systemic corticosteroid therapy (excluding topical, intranasal, inhaled, or other local routes) or any other form of immunosuppressive therapy within 7 days prior to the first study dose. The use of physiologic doses of corticosteroids (≤10 mg/day prednisone or equivalent) is permitted.
8. Severe hepatic or renal insufficiency.
9. Presence of any severe or uncontrolled systemic disease, including but not limited to:

   * Clinically significant, poorly controlled resting ECG abnormalities (e.g., complete left bundle branch block, second-degree or higher atrioventricular block, ventricular arrhythmia, or atrial fibrillation).
   * Unstable angina, congestive heart failure (New York Heart Association (NYHA) Class ≥ II).
   * Myocardial infarction within 6 months prior to randomization.
   * History of esophageal or gastric variceal bleeding within 6 months prior to enrollment.
   * Poorly controlled hypertension (systolic blood pressure >140 mmHg and/or diastolic blood pressure >90 mmHg).
   * History of non-infectious pneumonitis requiring corticosteroid treatment within 1 year prior to the first dose, or current clinically active interstitial lung disease.
   * Active tuberculosis.
   * Active or uncontrolled infection requiring systemic therapy.
   * Clinically active diverticulitis, intra-abdominal abscess, or gastrointestinal obstruction.
   * Decompensated liver disease, acute or chronic active hepatitis.
   * Unstable or active peptic ulcer disease, or patients with gastrointestinal bleeding.
   * Poorly controlled diabetes mellitus (fasting blood glucose >10 mmol/L).
   * Urinalysis indicating urine protein ≥ ++ and confirmed 24-hour urine protein quantification >1.0 g.
   * Uncontrolled hypercalcemia (>1.5 mmol/L ionized calcium, or calcium >12 mg/dL, or corrected serum calcium > ULN), or symptomatic hypercalcemia requiring continued bisphosphonate therapy.
   * Non-healing wound(s) or fracture(s).
   * Psychiatric disorder that compromises the ability to comply with the treatment protocol.
10. Female subjects who are pregnant or breastfeeding.
11. Assessed by the investigator as being unable or unwilling to comply with the requirements of the study protocol.
12. Known allergy to any of the study drug(s) used in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | Through out the study (up to 3 years)
  ORR was assessed by investigators per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
Progression-free Survival(PFS) | up to 3 years
  In treated subjects, the time from first recording to tumor progression (based on RECIST 1.1 and mRECIST) or death from any cause.

SECONDARY OUTCOMES:
Overall Survival(OS) | Up to 3 years
Adverse event | From the date of each patient's enrollment until 30 days (±7 days) after the last dose of study drug or until the initiation of new anti-tumor therapy, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Shen, Principal Investigator — Eastern Hepatobiliary Surgery Hospital

IPD SHARING:
Plan to Share IPD: No